CLINICAL TRIAL: NCT00783705
Title: Phase IIb Randomized Comparative Study of the Efficacy and Safety of Myo-inositol Versus Placebo in Smokers With Bronchial Dysplasia
Brief Title: Inositol in Preventing Lung Cancer in Current or Former Smokers With Bronchial Dysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00839; NCI-2009-00839 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000617846; MAY06-8-01 (Other: Mayo Clinic); MAY06-8-01 (Other: DCP); P30CA015083 (NIH)
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Non-small Cell Lung Cancer; Squamous Lung Dysplasia
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Inositol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (inositol) (Experimental): Patients receive oral inositol once daily for 2 weeks and then twice daily for up to 6 months in the absence of unacceptable toxicity.
  Interventions: Drug: inositol
- Arm II (placebo) (Experimental): Patients receive oral placebo once daily for 2 weeks and then twice daily for up to 6 months in the absence of unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II (placebo)
Drug: inositol — Given orally
  Other Names: myo-inositol
  Arms: Arm I (inositol)

SUMMARY:
This randomized phase II trial is studying inositol to see how well it works compared with a placebo in preventing lung cancer in current or former smokers with bronchial dysplasia. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of inositol may prevent lung cancer. It is not yet known whether inositol is more effective than a placebo in preventing lung cancer in smokers with bronchial dysplasia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of myo-inositol (inositol) 9 grams by mouth twice a day for 6 months versus placebo to revert bronchial dysplasia in current/former smokers with or without curatively treated Stage 0/I non-small cell lung cancer.

SECONDARY OBJECTIVES:

I. To further define the mechanism(s) of action of pharmacological doses of myo-inositol as a lung cancer chemopreventive agent by evaluating changes in: the number of dysplastic lesions, Ki-67, caspase-3, peroxisome proliferator-activated receptor (PPAR) gamma, cyclin D1, cyclin E and vascular endothelial growth factor (VEGF) immunostaining in bronchial biopsies; gene expression analysis of ribonucleic acid (RNA) from bronchial brush cells; and changes in inflammatory biomarkers (C-reactive protein [CRP], monocyte chemotactic protein-1 [MCP-1], myeloid progenitor inhibitory factor-1 [MPIF-1] and L-Selectin) levels in bronchoalveolar lavage (BAL) and plasma before and after treatment.

II. To collect additional safety and adverse event profiles of participants enrolled in both intervention arms. III. To establish a biospecimen repository archive for future correlative studies.

OUTLINE: Patients are stratified according to smoking status (current vs former), prior lung cancer (yes vs no), and number of dysplastic lesions at baseline (1 vs > 1). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral inositol once daily for 2 weeks and then twice daily for up to 6 months in the absence of unacceptable toxicity.

ARM II: Patients receive oral placebo once daily for 2 weeks and then twice daily for up to 6 months in the absence of unacceptable toxicity.

Patients undergo white light and autofluorescence bronchoscopy with bronchoalveolar lavage, bronchial brushings, and biopsies as well as optical coherence tomography imaging and blood sample collection at baseline and after completion of study treatment. Samples are analyzed for tissue biomarkers (e.g., PPAR gamma, Ki-67, caspase-3, cyclin D1, cyclin E, and VEGF) by immunohistochemistry (IHC); cytokine levels (e.g., CRP, MCP-1, MPIF-1, and L-selectin) by ELISA; and gene expression profiles of RNA by microarray.

After completion of study treatment, patients are followed within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed bronchial dysplasia in ≥ 1 site AND meets one of the following criteria:

  * Current or former smoker with ≥ a 30 pack-year smoking history and no history of lung cancer
  * Stage 0 or I non-small cell lung cancer (NSCLC) curatively treated by surgery (local ablation or resection), adjuvant chemotherapy, or radiotherapy with a ≥ 30 pack-year smoking history

    * At least 6 months since prior surgery, adjuvant chemotherapy, or radiotherapy
* No current evidence of lung cancer by CT scan

  * No non-calcified lung nodules ≥ 10 mm diameter on spiral CT scan unless cancer is ruled out by PET/CT scan or by biopsy
* ECOG performance status 0-1
* Hemoglobin normal
* Leukocyte count ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 1.5 times ULN
* ALT and AST ≤ 1.5 times ULN
* BUN ≤ 1.5 times ULN
* Chloride ≤ 1.5 times ULN
* Total CO_2 ≤ 1.5 times ULN
* Sodium ≤ 1.5 times ULN
* Calcium ≤ 1.5 times ULN
* Potassium ≤ 1.5 times ULN
* Phosphorus ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 30mL/min
* Fasting blood glucose normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No cancer within the past 3 years except stage 0 or I NSCLC, nonmelanomatous skin cancer, localized prostate cancer, carcinoma in situ of the cervix, or superficial bladder cancer that was treated > 6 months ago
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Severe chronic obstructive pulmonary disease requiring supplemental oxygen
  * Uncontrolled hypertension
  * Psychiatric illness or social situation that would limit compliance with study requirements
* No schizophrenia or bipolar disorder
* No diabetes
* No requirement for supplemental oxygen (continuous or intermittent)
* SaO_2 ≥ 90% on room air
* No history of allergic reactions attributed to inositol
* No history of allergies to any ingredient in the study agent or placebo
* No other concurrent investigational agents
* At least 7 days since prior anticoagulant use (e.g., coumadin or heparin)
* More than 6 months since prior participation in another chemoprevention clinical trial
* No prior pneumonectomy
* No prior solid organ transplantation
* No concurrent lithium, carbamazepine, or valproate
* No concurrent use of other natural health products containing inositol

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Limburg, Principal Investigator — Mayo Clinic
Locations (4):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - Albuquerque Veterans Administration Medical Center, Albuquerque, New Mexico
- BCCA-Vancouver Cancer Centre, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 448 subjects were pre-registered through 3 Cancer Prevention Network (CPN) member organizations from 2008 to 2013.
Pre-assignment Details: 363 subjects were excluded from pre-assignment: 342 ineligible via bronchoscopy, 3 participant decision, 13 lab values out of range, 1 screening time line issue and 4 suspicious of cancer.
Groups:
- Arm A (Myo-inositol): Patients receive oral inositol once daily for 2 weeks and then twice daily for up to 6 months in the absence of unacceptable toxicity.
- Arm B (Placebo): Patients receive oral placebo once daily for 2 weeks and then twice daily for up to 6 months in the absence of unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Started | 44 | 41
Completed | 38 | 36
Not Completed | 6 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo) | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Continuous [Median (Full Range); unit: years] | 58.5 [45.0 to 75.0] | 58.0 [46.0 to 79.0] | 58.0 [45.0 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 34 | 28 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 42 | 38 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
  Canada | 36 | 33 | 69
Body Mass Index, kg/m^2 [Median (Full Range); unit: kg/m^2] | 27.2 [21.1 to 36.3] | 26.0 [21.0 to 35.2] | 26.5 [21.0 to 36.3]
Smoking Status [Number; unit: participants]
  Current | 27 | 26 | 53
  Former | 17 | 15 | 32
Prior NSAID (nonsteroidal anti-inflammatory drugs) Use [Number; unit: participants]
  No | 28 | 29 | 57
  Yes | 16 | 12 | 28
Alcohol Intake [Number; unit: participants]
  1 or fewer drinks per day | 27 | 11 | 38
  2-3 drinks per day | 7 | 13 | 20
  4 or more drinks per day | 1 | 4 | 5
  None | 9 | 13 | 22
Dysplastic Lesions Identified [Number; unit: participants]
  1 Dysplastic lesion | 22 | 19 | 41
  >1 Dysplastic lesions | 22 | 22 | 44
Mucosal Biopsies Obtained [Median (Full Range); unit: biopsies] | 6.0 [1.0 to 14.0] | 7.0 [1.0 to 14.0] | 7.0 [1.0 to 14.0]
Most Advanced Histology [Number; unit: participants]
  Mild dysplasia | 15 | 13 | 28
  Moderate dysplasia | 28 | 22 | 50
  Severe dysplasia | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response Determined by Change in the Histologic Grade of Bronchial Dysplasia as Measured by Mucosal Biopsy Samples on Participant-specific Analysis.
Description: The definitions of responses are:
  Complete response: regression of all dysplastic lesion (DL) found at baseline to lesions that were no worse than hyperplasia and no new DL that were mild dysplasia or worse; Partial response: regression of some but not all of the DL with no new lesions that are mild dysplasia or worse; Progressive disease: progression of one or more sites by two or more grades or new DL that were mild dysplasia or worse; Stable disease: no complete response, partial response or progression.
Time Frame: From baseline up to 6 months
Population: The analysis population included the participants who received study intervention and completed both the pre- and post-intervention bronchoscopy.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
percentage of participants
  Complete response | 26.3 | 13.9
  Partial response | 10.5 | 16.7
  Stable disease | 15.8 | 36.1
  Progressive disease | 47.4 | 33.3

2. Primary Outcome: Percentage of Participants With Response Determined by Change in the Histologic Grade of Bronchial Dysplasia as Measured by Mucosal Biopsy Samples on Lesion-specific Analysis.
Description: The definitions of responses are:
  Complete response: the regression of a dysplastic lesion (DL) of any grade to one classified as being hyperplastic/normal; Progressive disease: appearance of lesions that were classified as mild dysplasia or worse; Stable disease: lesions that are not classified as complete response or progressive disease
Time Frame: From baseline up to 6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
percentage of participants
  Complete response | 10.2 | 7.4
  Stable disease | 15.9 | 22.6
  Progressive disease | 12.5 | 10.3
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Generalized estimating equation model on lesions (progressive disease vs. complete response/stable disease) was used to account for intra-patient correlation in the lesion-specific analysis; Test type: Superiority or Other; p = 0.39, Generalized estimating equation model; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.7 to 3.0]

3. Secondary Outcome: Percent Change in the Number of Bronchial Dysplastic Lesions Before and After Treatment
Description: The change in the number of bronchial dysplastic lesions is defined as disappearance or appearance of lesions.
Time Frame: From baseline up to 6 months
Population: The analysis population included the participants who received study intervention and completed both the pre- and post-intervention bronchoscopy with lesions biopsied.
Measure: Mean (Standard Deviation); unit: percentage change in number of lesions
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
percentage change in number of lesions | -53.5 (116.1) | -50.0 (115.8)

4. Secondary Outcome: Mean Percent Change in Ki-67 Expression Level in the Bronchial Biopsies With Dysplasia
Time Frame: From baseline up to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of Ki67 expression level
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 33 | 32
percentage of Ki67 expression level | -22.8 (105.3) | -6.2 (98.7)

5. Secondary Outcome: Change in Gene Expression Profiles of RNA in Bronchial Brush Cell Samples as Assessed by Microarray
Time Frame: From baseline up to 6 months
Population: Data were not collected due to a study team decision not to analyze this endpoint.
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Inflammatory Biomarkers Levels (CC-16) in Bronchoalveolar Lavage Samples as Assessed by Enzyme-linked Immunoassay (ELISA)
Description: The biomarkers that were examined were: 1) pro-inflammatory proteins: C-reactive protein (CRP, R&D Systems), interleukin-6 (IL-6, R&D Systems), and CCL-2 (R&D Systems); 2) oxidant/antioxidants: myeloperoxidase (MPO, R&D Systems), nitrotyrosine (Hycult Biotech) and glutathione (Millipore-Calbiochem); and 3) pneumoproteins: Clara cell protein-16 (CC-16, Biovendor), surfactant protein-D (SFTPD, R&D Systems) and CC18 (R&D Systems).
Time Frame: From baseline up to 6 months
Population: The analysis population included the participants who received study intervention and completed both the pre- and post-intervention bronchoscopy with bronchoalveolar lavage samples available
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
ng/mL | -66.96 [-127.56 to 52.26] | -54.32 [-144.65 to 140.84]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker CC-16 level between arms; Test type: Superiority or Other; p = 0.10, Wilcoxon Rank-Sum

7. Secondary Outcome: Change in Inflammatory Biomarkers Levels (IL-6) in Bronchoalveolar Lavage Samples as Assessed by Enzyme-linked Immunoassay (ELISA)
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
pg/mL | -0.68 [-2.78 to 0.34] | -0.27 [-1.54 to 1.89]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker IL-6 level between arms; Test type: Superiority or Other; p = 0.03, Wilcoxon Rank-Sum

8. Secondary Outcome: Change in Inflammatory Biomarkers Levels (CCL-2) in Bronchoalveolar Lavage Samples as Assessed by Enzyme-linked Immunoassay (ELISA)
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
pg/mL | -9.25 [-44.32 to 8.62] | 9.41 [-52.58 to 54.6]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker CCL-2 level between arms; Test type: Superiority or Other; p = 0.58, Wilcoxon Rank-Sum

9. Secondary Outcome: Change in Inflammatory Biomarkers Levels (MPO) in Bronchoalveolar Lavage Samples as Assessed by Enzyme-linked Immunoassay (ELISA)
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
ng/mL | -3.46 [-8.17 to 2.77] | -1.15 [-8.43 to 1.21]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker MPO level between arms; Test type: Superiority or Other; p = 0.06, Wilcoxon Rank-Sum

10. Secondary Outcome: Change in Inflammatory Biomarkers Levels (CC18) in Bronchoalveolar Lavage Samples as Assessed by Enzyme-linked Immunoassay (ELISA)
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
ng/mL | -121.47 [-1234.7 to 1122.9] | 10.70 [-684.95 to 683.25]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker CC18 level between arms; Test type: Superiority or Other; p = 0.63, Wilcoxon Rank-Sum

11. Secondary Outcome: Change in Inflammatory Biomarkers Levels (SFTPD) in Bronchoalveolar Lavage Samples as Assessed by Enzyme-linked Immunoassay (ELISA)
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
ng/mL | -12.39 [-47.12 to 5.72] | 7.21 [-7.62 to 23.79]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker SFTPD level between arms; Test type: Superiority or Other; p = 0.22, Wilcoxon Rank-Sum

12. Secondary Outcome: Change in Inflammatory Biomarkers Levels (Total Glutathione) in Bronchoalveolar Lavage Samples as Assessed by Enzyme-linked Immunoassay (ELISA)
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
umol/L | -0.25 [-1.98 to 0.48] | -0.56 [-1.13 to 0.33]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker Total Glutathione level between arms; Test type: Superiority or Other; p = 0.06, Wilcoxon Rank-Sum

13. Secondary Outcome: Change in Inflammatory Biomarkers Levels (CC-16) in Plasma Samples as Assessed by ELISA
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: The analysis population included the participants who received study intervention and completed both the pre- and post-intervention bronchoscopy with plasma samples available
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
ng/mL | -0.08 [-0.82 to 0.92] | -0.58 [-1.71 to 0.19]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker CC-16 level between arms; Test type: Superiority or Other; p = 0.35, Wilcoxon Rank-Sum

14. Secondary Outcome: Change in Inflammatory Biomarkers Levels (CRP) in Plasma Samples as Assessed by ELISA
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
ng/mL | 161.18 [-248.55 to 744.31] | -74.11 [-752.24 to 412.33]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker CRP level between arms; Test type: Superiority or Other; p = 0.80, Wilcoxon Rank-Sum

15. Secondary Outcome: Change in Inflammatory Biomarkers Levels (IL-6) in Plasma Samples as Assessed by ELISA
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
pg/mL | 0.06 [-0.74 to 0.46] | 0.01 [-0.55 to 0.73]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker IL-6 level between arms; Test type: Superiority or Other; p = 0.22, Wilcoxon Rank-Sum

16. Secondary Outcome: Change in Inflammatory Biomarkers Levels (CCL-2) in Plasma Samples as Assessed by ELISA
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
pg/mL | 2.19 [-35.08 to 29.56] | 9.08 [-5.53 to 44.08]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker CCL-2 level between arms; Test type: Superiority or Other; p = 0.74, Wilcoxon Rank-Sum

17. Secondary Outcome: Change in Inflammatory Biomarkers Levels (MPO) in Plasma Samples as Assessed by ELISA
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
ng/mL | 0.20 [-2.05 to 2.17] | 0.09 [-1.57 to 4.42]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker MPO level between arms; Test type: Superiority or Other; p = 0.55, Wilcoxon Rank-Sum

18. Secondary Outcome: Change in Inflammatory Biomarkers Levels (Nitrotyrosine) in Plasma Samples as Assessed by ELISA
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
mmol/L | 0.77 [-2.84 to 4.68] | 0.88 [-1.7 to 4]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker Nitrotyrosine level between arms; Test type: Superiority or Other; p = 0.91, Wilcoxon Rank-Sum

19. Secondary Outcome: Change in Inflammatory Biomarkers Levels (CC18) in Plasma Samples as Assessed by ELISA
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
ng/mL | 1.50 [-0.6 to 3.19] | -0.16 [-2.42 to 0.88]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker CC18 level between arms; Test type: Superiority or Other; p = 0.46, Wilcoxon Rank-Sum

20. Secondary Outcome: Change in Inflammatory Biomarkers Levels (SFTPD) in Plasma Samples as Assessed by ELISA
Description: as for outcome 6
Time Frame: From baseline up to 6 months
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Number analyzed (Participants) | 38 | 36
ng/mL | -0.28 [-0.93 to 1.51] | -0.22 [-1.26 to 2.22]
Statistical Analysis 1: Comparison: Arm A (Myo-inositol) vs Arm B (Placebo); Comparison of the median difference in biomarker SFTPD level between arms; Test type: Superiority or Other; p = 0.52, Wilcoxon Rank-Sum

ADVERSE EVENTS:
Description: Adverse events reported on all participants. The adverse events: cardiac disorders, blood disorders, gastrointestinal disorder and etc. which are simply repeating their organ system names were referred to other, specify category of the adverse events.
Arm/Group | Arm A (Myo-inositol) | Arm B (Placebo)
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/41
Other Adverse Events (participants affected / at risk) | 36/44 | 32/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Myo-inositol) (N=44) | Arm B (Placebo) (N=41)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Myo-inositol) (N=44) | Arm B (Placebo) (N=41)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 18 (26) | 9 (14)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 13 (16) | 3 (5)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (6) | 2 (2)
Chest pain (General disorders) | 5 (5) | 0 (0)
Chills (General disorders) | 5 (5) | 2 (2)
Fatigue (General disorders) | 6 (6) | 7 (10)
Fever (General disorders) | 4 (4) | 7 (8)
General symptom (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 2 (2)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Weight gain (Investigations) | 2 (2) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (7) | 4 (5)
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (3)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 6 (6)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 13 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (8)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (8)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (9)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less